CLINICAL TRIAL: NCT02483728
Title: Cutaneous and Systemic Reactions to Metal Implants: Utility of Patch Testing Prior and Post Placement of Metal Orthopedic Implants
Brief Title: Cutaneous and Systemic Reactions to Metal Implants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: NYU Langone Health (Other)
Collaborators: Smart Practice (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WUH 14318
Record Dates: First submitted 2015-06-17; First posted 2015-06-29 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Dermatitis, Allergic Contact
Keywords: Metal Allergy
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metal Allergy Hx +, Metal Patch Test + (Other): These are patients with a history of metal allergy who are patch test positive to metals (metal series, metal disc if available from manufacturer, bone cement components and topical antibiotics) prior to implantation of metal device.
  Interventions: Other: Patch Test
- Metal Allergy Hx +, Metal Patch Test - (Other): These are patients with a history of metal allergy who are patch test negative to metals (metal series, metal disc if available from manufacturer, bone cement components and topical antibiotics) prior to implantation of metal device.
  Interventions: Other: Patch Test

INTERVENTIONS:
Other: Patch Test — Patch testing is a technique used to diagnose an allergic skin disease called allergic contact dermatitis. It attempts to reproduce in small scale allergic reactions of the skin from things that come in contact with it.This is the standard of care to determine allergic contact dermatitis.

SUMMARY:
The purpose of this study is to evaluate if metal patch testing in metal allergic patients is useful for predicting the development of allergic skin disease or systemic symptoms in patients who recieve a metal orthopedic implant.

DETAILED DESCRIPTION:
This prospective cohort study will enroll patients with a history of metal allergy who require implantation of a metal orthopedic device. Patients will be followed for one year after surgery to determine if any symptoms including rash, itch, joint pain, joint swelling, and/or joint failure develop post implantation.

Patients will be recruited from two sites: (1) Divisions of Orthopedics and Allergy & Immunology, Winthrop University Hospital, and (2) Division of Immunology, and Allergy Section, University of Cincinnati Medical Center.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years with a history of metal allergy who require joint repair (hip, knee and/or shoulder)
2. Able to undergo patch testing

Exclusion Criteria

1. Patients on oral immunosuppressant medications within 4 weeks of patch testing or topical corticosteroids to the back within 1 week of patch testing
2. Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
The development of rash assessed via a patient and physician questionnaire asking to answer yes or no to the following questions: Do you have new onset of itchy rash above the implant site? Do you have new onset of generalized itchy rash? | Change from baseline physical exam prior to surgery (development of rash) at 4-6 weeks post date of surgery, 3 months post surgery, 6 months post surgery and one year post surgery.
  Type of rash that has developed: eczema above implant, generalized eczema, urticaria, vasculitis
The development of joint pain or joint swelling assessed via a patient and physician questionnaire asking to answer yes or no to the following questions: Do you have pain at the site of your implant? Does the patient have atypical joint swelling? | Change from baseline physical exam prior to surgery at 4-6 weeks post date of surgery, 3 months post surgery, 6 months post surgery and one year post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marcella Aquino, MD, Principal Investigator — NYU Winthrop Hospital
Locations (2):
- United States (2):
  - Winthrop University Hospital, Mineola, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio

REFERENCES:
- [Background] Pinson ML, Coop CA, Webb CN. Metal hypersensitivity in total joint arthroplasty. Ann Allergy Asthma Immunol. 2014 Aug;113(2):131-6. doi: 10.1016/j.anai.2014.05.012. Epub 2014 Jun 13. PMID 24934108